CLINICAL TRIAL: NCT05140213
Title: EVALUATION OF 30-DAY MORTALITY AFTER A VISIT TO THE LAPEYRONIE ADULT EMERGENCY DEPARTMENT OF THE CHU MONTPELLIER FOR SEPSIS OR SEPTIC SHOCK
Brief Title: A STUDY BEFORE/AFTER THE IMPLEMENTATION OF AN ANTI-INFECTIOUS PRESCRIPTION AID
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0685
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Sepsis; Septic Shock
Keywords: Adult patients; Probabilistic antibiotic therapy to be initiated
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 : Before: "Before" phase including 186 patients patients included before the implementation of the prescription support tool
  Interventions: Device: Anti-infectious prescription support tool
- Group 2 : After: "After" phase including 185 patients patients included after the implementation of the prescription support tool
  Interventions: Device: Anti-infectious prescription support tool

INTERVENTIONS:
Device: Anti-infectious prescription support tool — implementation of a pocket notebook with current anti-infectious recommendations in the emergency department Patients were kept under surveillance for at least one hour before discharge.
  Patients were discharged home with a 7 day supply of acetaminophen 1000 mg orally every 6 h, ketoprofen 100 mg, orally twice a day, and muscle relaxant as needed. Patients were instructed to take tramadol 50 mg, orally every 6h as needed for low back pain, in case of insufficient relief.

SUMMARY:
Anti-infective strategy is a major public health problem. This is a before-and-after study of an anti-infectious prescription tool with a comparison of mortality at 30 days (then 3 and 6 months) between the two inclusion phases of 6 months each.

ELIGIBILITY:
Inclusion criteria:

* Major patients
* Sepsis or septic shock
* Oral consent

Exclusion criteria:

* minor patients
* death before antibiotherapy
* care limitations
* pre-hospital antibiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with severe sepsis in the Montpellier emergency department
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Numbers of patient 30-day mortality | 30 day
  patient survival at 30 days

OTHER OUTCOMES:
Numbers of patient 90-day mortality | 90 days
  patient survival at 90 days
Numbers of patient 6 months mortality | 6 months
  patient survival at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamza GHOMRANI, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC